CLINICAL TRIAL: NCT00141128
Title: Measurement Of Urethral Function In Women With Stress Urinary Incontinence - Evaluation Of The Sensitivity Of Urethral Reflectometry Compared To Urethral Pressure Profilometry, Using [S,S]-Reboxetine To Detect Pharmacological Augmentation Of Urethral Pressure.
Brief Title: Evaluation Of A Novel Methodology In The Assessment Of Urethral Function Using SS-RBX.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A6061024
Record Dates: First submitted 2005-08-29; First posted 2005-09-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

INTERVENTIONS:
Drug: SS-RBX

SUMMARY:
SS-RBX will be used to evaluate pharmacodynamic changes in urethral function using a novel methodology

ELIGIBILITY:
Inclusion Criteria:

* Female
* Stress urinary incontinence

Exclusion Criteria:

* Bladder outflow obstruction
* Neurological disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-12; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To assess the utility of urethral reflectometry in the detection of pharmacologically induced pressure changes in the female urethra.

SECONDARY OUTCOMES:
To assess the effect of [S,S]-Reboxetine on urethral function in women with SUI.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Klarskov N, Scholfield D, Soma K, Darekar A, Mills I, Lose G. Measurement of urethral closure function in women with stress urinary incontinence. J Urol. 2009 Jun;181(6):2628-33; discussion 2633. doi: 10.1016/j.juro.2009.01.114. Epub 2009 Apr 16. PMID 19375093
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061024&StudyName=Evaluation+Of+A+Novel+Methodology+In+The+Assessment+Of+Urethral+Function+Using+SS%2DRBX%2E